CLINICAL TRIAL: NCT07287111
Title: Multi-Reader Multi-Case, Cross-Over, Retrospective Study to Evaluate the Effectiveness of CadAI-B Dx for Decision Support in Breast Ultrasound
Brief Title: Effectiveness of CadAI-B Dx for Decision Support in Breast Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BeamWorks Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: IP0014-US-CAB-I
Record Dates: First submitted 2025-12-11; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Retrospective, fully-crossed, Multi-Reader Multi-Case (MRMC) study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CadAI- Dx(AI) Unaided Reading (No Intervention): Readers evaluate each ultrasound image without access to AI assistance. Readers use only the provided radiological images and their professional clinical expertise to determine their final diagnosis and relevant findings
- CadAI-DX (AI)-aided Reading (Experimental): Readers have access to CadAI-B's decision-support outputs, which include a pixel-level heatmap (CadAI-Map), auto-segmented lesion boundary, BI-RADS lexicon descriptors, a suggested malignancy probability score (CadAI-Score), and BI-RADS category.
  Interventions: Device: CadAI-B Dx

INTERVENTIONS:
Device: CadAI-B Dx — CadAI-B Dx is a Software as a Medical Device (SaMD) designed to assist physicians by providing Computer-Aided Detection (CADe) and Diagnosis (CADx) capabilities in breast ultrasound interpretation. The software automatically processes the image to identify suspicious regions (Lesion Detection) and provides a quantitative malignancy score (CadAI-Score) mapped to a corresponding BI-RADS Category. It also analyzes lesion size and BI-RADS lexicon descriptors.
  Arms: CadAI-DX (AI)-aided Reading

SUMMARY:
This is a retrospective, fully-crossed, multi-reader, multi-case (MRMC) study to evaluate the effectiveness of 'CadAI-B Dx' (CadAI-B) for decision support in breast ultrasound. The study compares the diagnostic performance of readers interpreting breast ultrasound images with and without the aid of CadAI-B. A total of 797 patient cases will be included, comprising 350 cases with a confirmed diagnosis of malignancy and 447 cases with a confirmed benign diagnosis. Sixteen readers will participate in the study to evaluate the device.

DETAILED DESCRIPTION:
The study utilizes a crossover design where all readers independently review all cases. The control arm consists of a reading session where participating readers independently review cases without the assistance of the CadAI-B device (unaided reading). The experimental arm involves reading with CadAI-B assistance (AI-aided reading). To minimize potential bias, a washout period of four weeks will be maintained between the unassisted and assisted reading sessions for each reader. The primary hypothesis is that CadAI-B assistance significantly improves overall reader performance in breast ultrasound interpretation, as measured by the area under the Localization Receiver Operating Characteristic (LROC) curve (AULROC).

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 22 years or older at the time of the breast ultrasound examination.
2. Standard B-mode breast ultrasound images available for analysis.
3. Lesions must have a confirmed diagnosis based on one of the following reference standards:

3-1. Malignant Cases: Diagnosis of breast cancer confirmed through biopsy or surgery.

3-2. Benign Cases: Confirmed as benign through biopsy or surgical excision, or confirmed as having no evidence of malignancy for at least 2 years of follow-up.

Exclusion Criteria:

1. mages containing modes other than standard B-mode ultrasound, such as Doppler, elastography, or other annotations/overlays.
2. Patients who have breast implant(s).
3. Patients suffering from significant breast trauma or mastitis at the time of the breast ultrasound examination.
4. Images of post-surgical resection sites.
5. Images where multiple lesions are present within a single 2D ultrasound image

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 797 (Actual)
Dates: Start 2025-08-30 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Area Under the Localization Receiver Operating Characteristic (LROC) Curve (AULROC) | Through study completion, approximately 2 months
  The difference in reader performance between the unaided and AI-aided sessions in breast ultrasound interpretation. LROC reflects both detection accuracy and localization precision. The primary hypothesis is that the mean AULROC of all readers for the AI-aided reading mode is greater than that for the unaided reading mode.

SECONDARY OUTCOMES:
Sensitivity | Through study completion, approximately 2 months
  Comparison of the average sensitivity of the readers between the unaided and AI-aided sessions.
Positive Predictive Value (PPV) | Through study completion, approximately 2 months
  Comparison of PPV between unaided and AI-aided sessions. The PPV will be adjusted for disease prevalence in the target population to reflect real-world clinical practice.
Negative Predictive Value (NPV) | Through study completion, approximately 2 months
  Comparison of NPV between unaided and AI-aided sessions. The NPV will be adjusted for disease prevalence in the target population.
Inter-reader Agreement | Through study completion, approximately 2 months
  Evaluation of the consistency of interpretations among different readers. Inter-reader agreement for BI-RADS category and descriptors assignments will be compared between sessions using Kappa statistics.
Reading Time | Through study completion, approximately 2 months
  Comparison of the average reading time per case between the unaided and AI-aided sessions to assess if the AI system improves the efficiency of interpretation.
AI-Ground Truth Agreement | Through study completion, approximately 2 months
  Assessment of the agreement between the AI system's outputs and the ground truth. This includes agreement on BI-RADS categories and descriptors (using Kappa statistics) and lesion size measurements (using Intraclass Correlation Coefficient).

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
ndividual participant data will not be shared to protect proprietary information and subject confidentiality.